CLINICAL TRIAL: NCT00728208
Title: A Placebo-controlled, Single-blind, Randomised, Parallel Group, 28-day Repeat Dose Study to Investigate the Tolerability, Safety and Steady State Pharmacokinetics of GSK372475 in Healthy Young and Elderly, Male and Female Subjects
Brief Title: GSK372475 PK Study in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 105467
Record Dates: First submitted 2008-07-31; First posted 2008-08-05 (Estimated); Last update posted 2017-07-13 (Actual); Status verified 2017-07

CONDITIONS: Depressive Disorder
Keywords: Young; Elderly; Randomised; GSK372475
MeSH Terms: conditions — Depressive Disorder | interventions — GSK372475

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (1):
- GSK372475 (Experimental): Drug
  Interventions: Drug: GSK372475

INTERVENTIONS:
Drug: GSK372475 — 1.5mg for 28 days

SUMMARY:
This study will consist of 4 parallel cohorts of healthy volunteers (elderly male, elderly female, young male and young female). Subjects will receive either GSK372475 1.5mg or placebo for 28 days.

ELIGIBILITY:
Inclusion Criteria:

* Healthy as determined by a responsible physician, based on a medical evaluation including medical and psychiatric history (including family history), full physical examination, laboratory tests and cardiac monitoring.
* Male or female between 18 and 45 years of age (young healthy population) and >65 years old (elderly population).
* A female subject is eligible to participate if she is of:
* Non-childbearing potential defined as pre-menopausal females with a documented tubal ligation or hysterectomy; or postmenopausal defined as 12 months of spontaneous amenorrhea
* Child-bearing potential and agrees to use of specific contraception methods. Use of oral contraception is permitted.
* BMI within the range 19 - 29 kg/m2 (inclusive).
* Capable of giving written informed consent, which includes compliance with the requirements and restrictions listed in the consent form.
* QTcB or QTcF < 450 msec; or QTc < 480 msec in subjects with Bundle Branch Block.
* Able to swallow and retain oral medication

Exclusion Criteria:

* A subject will not be eligible for inclusion in this study if any of the following criteria apply:
* Evidence or history of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular or other heart disease, glaucoma, diabetes, hepatic, neurologic (e.g. including but not limited to seizures, stroke, cerebrovascular disease or other brain conditions), or allergic disease (except for untreated, asymptomatic, seasonal allergies at time of dosing).
* Psychiatric illness currently or within the past year, or any lifetime history of bipolar disorder, major depressive disorder, anxiety disorder, schizophrenia or other psychotic disorder, or substance abuse or dependence (except past history of nicotine abuse/dependence).
* Subjects who, in the investigator's judgment, pose a suicidal or homicidal risk, or any subject with a history of suicidal or homicidal attempts or behaviour.
* The subject has a positive pre-study drug/alcohol screen. A minimum list of drugs that will be screened for include amphetamines, barbiturates, cocaine, opiates, cannabinoids and benzodiazepines.
* A positive pre-study Hepatitis B surface antigen or positive Hepatitis C antibody result within 3 months of screening (with the exception of phase I hepatic impairment studies, oncology studies, hepatitis, hepatic fibrosis, or HIV studies).
* A positive test for HIV antibody.
* History of regular alcohol consumption within 6 months of the study defined as:
* an average weekly intake of greater than 21 units or an average daily intake of greater than 3 units (males), or defined as an average weekly intake of greater than 14 units or an average daily intake of greater than 2 units (females). One unit is equivalent to a half-pint (220mL) of beer or 1 (25ml) measure of spirits or 1 glass (125ml) of wine.
* The subject has participated in a clinical trial and has received an investigational product within the following time period prior to the first dosing day in the current study: 60 days i.e. 5 half-lives.
* Exposure to more than four new chemical entities within 12 months prior to the first dosing day.
* Use of prescription or non-prescription drugs, including vitamins, herbal and dietary supplements (including St John's Wort) within 7 days (or 14 days if the drug is a potential enzyme inducer) or 5 half-lives (whichever is longer) prior to the first dose of study medication, unless in the opinion of the Investigator and GSK Medical Monitor the medication will not interfere with the study procedures or compromise subject safety.
* History of sensitivity to any of the study medications, or components thereof or a history of drug or other allergy that, in the opinion of the investigator or GSK Medical Monitor, contraindicates their participation.
* Where participation in the study would result in donation of blood or blood products in excess of 500 mL within a 56 day period.
* Pregnant females as determined by positive serum or urine hCG test at screening or prior to dosing.
* Lactating females.
* Administration of a monoamine oxidase inhibitor (MAOI) within 30 days prior to Study Day 1, or anticipated use within 12 weeks following the last dose of study drug.
* Unwillingness or inability to follow the procedures outlined in the protocol.
* History of sensitivity to heparin or heparin-induced thrombocytopenia.
* Consumption of grapefruit juice or grapefruit or cruciferous vegetables (e.g. broccoli, Brussels sprouts, cabbage, cauliflower, chard, kale, mustard greens, rutabagas and turnips) and charbroiled foods within 7 days prior to first dose of study medication until follow-up.
* Controlled or uncontrolled hypertension, or systolic blood pressure ≥140 mmHg or diastolic blood pressure ≥90 mmHg at screening or prior to the first dose of study medication.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2008-07-28 (Actual); Primary Completion 2008-12-29 (Actual); Study Completion 2008-12-29 (Actual)

PRIMARY OUTCOMES:
Main pharmacokinetic parameters after single and repeat administration: Cmax, tmax, AUC(0-t), AUC(0-tau), Ctau and Ro. | pre-dose to 24 hours post dose

SECONDARY OUTCOMES:
Safety and tolerability endpoints, including adverse events (AEs), vital signs, electrocardiograms (ECGs) and clinical laboratory tests. | from dosing to follow-up

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Berlin, Germany

REFERENCES:
- See also: Results for study 105467 can be found on the GSK Clinical Study Register. — https://www.gsk-clinicalstudyregister.com/study/105467?search=study&search_terms=105467#rs